CLINICAL TRIAL: NCT04226963
Title: A Naturalistic Study of Ketamine for Treatment Resistant Mood Disorders: Gdansk Depression Ketamine Project
Brief Title: A Naturalistic Study of Ketamine for Treatment Resistant Mood Disorders
Acronym: GDKet
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Maria Galuszko-Wegielnik, Principal Investigator, Clinical doctor, Medical University of Gdansk
Other Study IDs: NKBBN/172-674/2019
Record Dates: First submitted 2020-01-02; First posted 2020-01-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Treatment Resistant Depression; Bipolar Depression; Ketamine; Major Depressive Disorder
Keywords: treatment resistant depression; bipolar depression; ketamine; multiple series; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Bipolar Disorder; Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ketamine — Ketamine will be infused (slow IV infusions of ketamine (0.5 mg/kg) over 40 minutes) twice weekly over a period of 4 weeks) Ketamine will be given in intranasal spray twice weekly over a period of 4 weeks Ketamine will be given orally (solution 2.0mg/kg, 2.5mg/kg) twice weekly over a period of 4 weeks.

SUMMARY:
This study aims to openly test the long-term safety, tolerability and effectiveness of repeated administration of IV, nasal spray and oral ketamine for treatment-resistant mood disorders.

DETAILED DESCRIPTION:
Current pharmacological treatments for depression prove unsatisfactory efficacy with a proportion of subjects demonstrating treatment-resistant depression (TRD). The observation applies both to major depressive disorder (MDD) as well as bipolar I depression. There is growing evidence that the glutamatergic system plays a role in the pathophysiology and treatment of depression. Discovery of rapid, although transient antidepressant effect of ketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist used in a single sub-anaesthetic intravenous dose in unipolar, bipolar and treatment-resistant patients provides evidence for a glutamatergic antidepressant. Subsequent studies confirmed this effect in repeated doses. Further research demonstrated that repeated ketamine infusions result in sustainable antidepressant effect with both, twice-weekly and thrice-weekly administration schedules. However, the worsening of depression may occur after infusions are completed. Given the risk of relapses, there is a definite need for the development of new strategies to maintain the beneficial effects of ketamine treatment. In the present study, the investigators aim to openly assess the safety, tolerability, and effectiveness of repeated, individually tailored IV, nasal spray and oral ketamine for treatment-resistant mood disorders. The investigators intend to explore questions regarding optimal dose, treatment frequency and duration.

ELIGIBILITY:
Inclusion Criteria:

1. Major depressive disorder (MDD) or bipolar disorder (BD) diagnosis as provided by DSM-5 criteria
2. TRD defined as the patient does not reach remission within the 8 week trial of an antidepressant or combination at a therapeutic dose of at least two trials of first-line evidence-based treatments and/or electroconvulsive therapy (ECT)

Exclusion Criteria:

1. Pregnancy and lactation
2. Hypersensitivity to ketamine
3. Uncontrolled hypertension
4. Other uncontrolled somatic diseases that may impact safety per investigators judgement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with TRD referred to the tertiary-reference unit for mood disorders
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events assessed by Clinical-Administered Dissociative Symptoms Scale (CADSS) | Baseline through week 5
  Incidence of adverse events will be assessed by Clinician-Administered Dissociative Symptoms Scale (change from baseline to each measure). Higher values represent a worse severity, but not necessarily outcome. The Clinical-Administered Dissociative Symptoms Scale has 23-items based on dissociative symptoms during the assessment. Each item is scored 0 (normal) to 4 (severe symptoms) with overall score ranges from 0 (normal) to 92 (severe symptoms). Total number of assessments:18 times
Incidence of adverse events assessed by 4-items positive symptoms subscale of Brief Psychiatric Rating Scale (BPRS) | Baseline through week 5
  Incidence of adverse events will be assessed by 4-items positive symptoms subscale of Brief Psychiatric Rating Scale (change from baseline to each measure). Higher values represent a worse severity but not necessarily outcome. The 4-item positive symptoms subscale of Brief Psychiatric Rating Scale has 4-items based on conceptual disorganization, suspiciousness, hallucination and unusual thought content. Each item is scored 0 (normal) to 6 (severe symptoms) with overall score ranges from 0 (normal) to 24 (severe symptoms). Total number of assessments:18 times
Incidence of adverse events assessed by body temperature (oral measurements) | Baseline through week 5
  Incidence of adverse events assessed by body temperature (oral measurement) in Celsius degree - change from baseline to each measure. A normal range is from 36.2 to 38.0 Celsius degrees; measurements beyond those ranges are clinically significant. The total number of measurements: 44 times
Incidence of adverse events assessed by blood pressure | Baseline through week 5
  Incidence of adverse events assessed by blood pressure (after the participant has rested for at least 5 minutes) in mmHg - change from baseline to each measure. A normal range for systolic blood pressure is from 90 to 140 mmHg, for diastolic blood pressure is from 50 to 90 mmHg; measurements beyond those ranges are clinically significant. The total number of measurements: 44 times
Incidence of adverse events assessed by respiration rate | Baseline through week 5
  Incidence of adverse events assessed by respiration rate in a breath number per minute - change from baseline to each measure. A normal range for respiration is from 12 to 16 breaths per minute; measurements beyond those ranges are clinically significant. The total number of measurements: 44 times
Incidence of adverse events assessed by pulse | Baseline through week 5
  Incidence of adverse events assessed by pulse (beats per minute [bpm]) - change from baseline to each measure. A normal range for pulse is from 60 to 90 bpm; measurements beyond those ranges are clinically significant. The total number of measurements: 44 times
Incidence of adverse events assessed by blood oxygen saturation | Baseline through week 5
  Incidence of adverse events assessed by blood oxygen saturation in percentage - change from baseline to each measure. A normal range for blood oxygen saturation is from 95 to 100 percentage; measurements under 95% are clinically significant. The total number of measurements: 44 times
Incidence of adverse events assessed by weight | Baseline and week 5
  Incidence of adverse events assessed by weight in kilograms- change from baseline to each measure. Gain weight for 7% baseline weight is clinically significant. Total numbers of assessments: 2. Weight and height will be combined to report BMI in kg/m^2
Incidence of adverse events assessed by height | Baseline
  Incidence of adverse events assessed by height in meters. Total numbers of assessments: 1. Weight in kilograms and height in meters will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Change in severity of depression symptoms assessed by Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline through week 5
  Change in severity of depression symptoms from baseline to each measure. Higher values represent a worse severity, but not necessarily outcome. The MADRS has 10-items which are based on mood symptoms over the past 7 days. Each item is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Medical University of Gdańsk, Gdansk, Poland

REFERENCES:
- [Derived] Kachlik Z, Cubala WJ, Walaszek M, Pastuszak M, Pastuszak K, Kwasny A. Nonresponse to Ketamine in Treatment-Resistant Bipolar Depression. Neuropsychopharmacol Rep. 2025 Sep;45(3):e70038. doi: 10.1002/npr2.70038. PMID 40879542
- [Derived] Wlodarczyk A, Cubala WJ, Galuszko-Wegielnik M, Szarmach J. Dissociative symptoms with intravenous ketamine in treatment-resistant depression exploratory observational study. Medicine (Baltimore). 2021 Jul 23;100(29):e26769. doi: 10.1097/MD.0000000000026769. PMID 34398056
- [Derived] Wlodarczyk A, Cubala WJ, Galuszko-Wegielnik M, Szarmach J. Central nervous system-related safety and tolerability of add-on ketamine to antidepressant medication in treatment-resistant depression: focus on the unique safety profile of bipolar depression. Ther Adv Psychopharmacol. 2021 May 19;11:20451253211011021. doi: 10.1177/20451253211011021. eCollection 2021. PMID 34046159